CLINICAL TRIAL: NCT03925844
Title: Cardiovascular Risk in People Older Than 55 Years and Cognitive Performance at 5 Years: an Estimation Model Based on Spanish Population. NEDICES-2-RISK Study.
Brief Title: Cardiovascular Risk in People Older Than 55 Years and Cognitive Performance at 5 Years
Acronym: NEDICES2RISK
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Responsible Party: Principal Investigator, Ester Tapias Merino, Clinical researcher, Gerencia de Atención Primaria, Madrid
Other Study IDs: PI18/00522
Record Dates: First submitted 2019-03-24; First posted 2019-04-24 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Risk Factor, Cardiovascular; Cognitive Decline
Keywords: Cardiovascular risk prediction models; Framingham risk function; FRESCO risk function; risk function; cognitive aging; prevention
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Classification according to the cardiovascular risk — All patients are cognitively assessed at the beginning of the study and their cardiovascular risk is calculated. After 5 years of follow-up, patients are re-evaluated cognitively and their cardiovascular risk is recalculated.

SUMMARY:
This study assesses whether people's cardiovascular risk influences cognitive performance in later years. To do this, the cardiovascular risk and cognitive performance of each patient will be evaluated at the beginning of the study and 5 years later.

ELIGIBILITY:
Inclusion Criteria:

* population aged 55 to 74 years from NEDICES 2 study
* to have signed informed consent
* to have done the neuropsicological assessment

Exclusion Criteria:

* to have a dementia diagnosis at baseline.

Ages: 55 Years to 74 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population comes from the cohort NEDICES 2. NEDICES 2 population comes from primary care physician´s lists.
Sampling Method: Probability Sample
Enrollment: 965 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change in the 37-item versión of the Mini-Mental State Examination score | Baseline and 5 years
  The 37 item Version of the Mini-Mental State Examination is a Spanish adapted version of the original MMSE by Folstein. It contains 37 items. Includes temporal and spatial orientation, memory, attention, calculus, language, object recognition, elementary commands and visuoconstructive capacity. The minimun score is 0 and the maximum score is 37 points. Higher values are considered a better outcome.
Change in the Clock-drawing test score | Baseline and 5 years
  The Clock-drawing test is a brief test that explores comprehension, concentration, visual memory and abstraction and visuoconstructive praxis. The subject is asked to draw a clock from memory on a blank sheet, including the numbers and hands at a fixed time. The minimum score is 0 and the maximum score is 4. Higher values are considered a better outcome. Performance time is recorded. A shorter time is considered a better outcome.
Change in the Center for Epidemiologic Studies Depression Scale (CES-D) score | Baseline and 5 years
  The Center for Epidemiologic Studies Depression Scale (CES-D) is a screening instrument for depression, self-administared, which records depressive symptoms and their different manifestations in the last 7 days and each symptom is classified in four frequency levels. The score ranges from 20 to 80. Higher values are considered a worse outcome.
Change in the Semantic verbal fluency test score | Baseline and 5 years
  The Semantic verbal fluency test evaluates semantic memory, executive and verbal planning capabilities. It is used a shorter version that evaluates the number of elements in a category (animals). There is a minimum score of 0, there is not a maximun score. Higher values are considered a better outcome.
Change in the Six-object memory recall test score | Baseline and 5 years
  The Six-Object Memory Recall Tests shows six sheets with common objects and explores object recognition, immediate recall and delayed memory after 5 minutes. Both, object recognition, inmediate recall and delayed memory have a scale ranging from 0 to 6.Therefore, the total score has a minimun score of 0 and a maximum score of 18 points. Higher values are considered a better outcome.
Change in the Mental Function Index score | Baseline and 5 years
  The Mental Function Index is a questionnaire that evaluates 11 instrumental activities of daily life and competencies in the home and occupational and social functioning that is administered to a family member or caregiver. It explores 11 sections, each one with three levels of functionality. The minimum score is 0 and the maximum score is 33. Higher values are considered a worse outcome.
Change in the Trail Making Test score | Baseline and 5 years
  The Trail Making Test is a visuomotor integration test from which is collected the score, the number of mistakes and the performance time. The score ranges from 1 to 20. Higher values are considered a better outcome. A shorter performance time and fewer mistakes are considered a better outcome.
Change in the Word accentuation test score | Baseline and 5 years
  The Word accentuation test is a verbal intelligence test in which the participant reads 30 unusual words that are shown to him without tildes and whose accentuation he has to do correctly. The score ranges from 0 to 30. Higher values are considered a better outcome.

SECONDARY OUTCOMES:
New cases of cancer during the 5-years follow-up | 5 years
  It will be recorded all new cases of cancer during the 5-years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ester Tapias-Merino, MD, Principal Investigator — Gerencia de Atención Primaria, Madrid
Locations (1):
- Gerencia Atencion Primaria, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Hernandez-Gallego J, Llamas-Velasco S, Bermejo-Pareja F, Vega S, Tapias-Merino E, Rodriguez-Sanchez E, Boycheva E, Serrano JI, Gil-Garcia JF, Trincado R, Sanchez-Rodrigo JV, Cacho J, Contador I, Garcia-Ptacek S, Sierra-Hidalgo F, Cubo E, Carro E, Villarejo-Galende A, Garcia Garcia-Patino R, Benito-Leon J. Neurological Disorders in Central Spain, Second Survey: Feasibility Pilot Observational Study. JMIR Res Protoc. 2019 Jan 10;8(1):e10941. doi: 10.2196/10941. PMID 30632964
- [Derived] Tapias-Merino E, De Hoyos-Alonso MDC, Contador-Castillo I, Rodriguez-Sanchez E, Sanz-Cuesta T, Becerro-Munoz CM, Hernandez-Gallego J, Vega-Quiroga S, Bermejo-Pareja F; NEDICES2-RISK Group. Cardiovascular risk in subjects over 55 years of age and cognitive performance after five years. NEDICES2-RISK study. Study protocol. PLoS One. 2022 Nov 28;17(11):e0274589. doi: 10.1371/journal.pone.0274589. eCollection 2022. PMID 36441718

DOCUMENTS (2):
  • Informed Consent Form (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT03925844/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT03925844/Prot_SAP_001.pdf